CLINICAL TRIAL: NCT06211114
Title: Study to Evaluate the Efficacy and Safety of Immune Checkpoint Inhibitors in Combination With Axitinib in Previously Treated Advanced Collecting Duct Carcinoma
Brief Title: Study to Evaluate the Efficacy and Safety of Immunotherapy With Axitinib in Advanced Collecting Duct Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, MD., Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FD-001-II-RCC
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Collecting Duct Carcinoma
Keywords: Immune Checkpoint Inhibitors; Axitinib
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-(L)1 inhibitor + Axitinib (Experimental): Immune Checkpoint Inhibitors in Combination With Axitinib
  Interventions: Drug: PD-(L)1 inhibitor; Drug: Axitinib

INTERVENTIONS:
Drug: PD-(L)1 inhibitor — Toripalimab 240mg or Tirelizumab 200mg or pembrolizumab 200mg intravenously every 3 weeks
Drug: Axitinib — axitinib 5mg orally twice daily

SUMMARY:
This is a phase II trial to evaluate the efficacy and safety of immune checkpoint inhibitors in combination with axitinib for previously treated advanced collecting duct carcinoma.

DETAILED DESCRIPTION:
Patients meeting specific inclusion and exclusion criteria will be enrolled in two stages, 8 patients in stage 1 and 22 patients in stage 2. Stage 2 will enroll if 1 or more patients exhibit a response at week 9 or later in stage 1 in the study. All enrolled patients will be treated with immune checkpoint inhibitors in combination with axitinib until disease progression. Efficacy will be assessed by tumor measurements using CT and MRI (when indicated) scans and physical exam at baseline, and scans and physical exam of all disease-involved areas every 9 weeks until progression. Safety will be assessed by periodic physical exams, clinical laboratory studies, and adverse events. All patients will have a follow-up visit 90 days following last study drug treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand and be willing to provide written informed consent.
2. Male or female with age ≥ 18 years and <80 years.
3. Have received prior systemic therapy after previous metastasis for collecting duct carcinoma, histologically confirmed diagnosis of unresectable, recurrent or metastatic collecting duct carcinoma.
4. Having at least one measurable disease per RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if re-progression has been demonstrated.
5. ECOG PS 0 or 1.
6. Adequate function of vital organs:

   6.1 Bone marrow function (without blood or blood products transfusion, without hematopoietic stimulating factor or other medication to improve blood cell count within 2 days prior to first dose of study drug): Absolute neutrophil count (ANC) ≥ 1.5×109/L. Platelets ≥ 100×109/L. Hemoglobin ≥ 9.0g/dL or ≥ 5.6mmol/L. 6.2 Renal function: Serum creatinine ≤ 1.5×ULN 6.3 Hepatic function:Serum total bilirubin ≤1.5×ULN or total bilirubin levels >1.5×ULN with direct bilirubin ≤ ULN. AST and ALT ≤2.5 × ULN, ≤5×ULN in those with hepatic metastasis.

   6.4 Endocrine function: Normal thyroid stimulating hormone, or abnormal TSH whilst normal FT3 and FT4.

   6.5 Coagulation function: International normalized ratio (INR) or prothrombin time (PT) ≤1.5×ULN, and activated partial thromboplastin time (aPTT) ≤1.5×ULN, Subjects receiving anticoagulant therapy (e.g., heparin or warfarin) may participate in the study with PT or APTT levels within the scope of the proposed therapy and monitored during study treatment.

   6.6 Left ventricular ejection fraction (LVEF) ≥ 50%.
7. Being willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
8. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first treatment dose. Female subjects of childbearing potential and male subjects whose partners are of childbearing potential must agree to use a highly effective methods of contraceptive throughout the study and for 180 days after the last dose of study therapy.

Exclusion Criteria: Exclusion criteria: Patients with any of the following conditions will not be included in the study:

1. Prior Anti-PD-1, PD-L1 or axitinib.
2. Has participated or is currently participating in a trial of investigational agent within 4 weeks prior to the first dose of study treatment, unless observational (non-interventional) clinical study or follow-up period of interventional study.
3. Had major surgery (judged by investigators) within 4 weeks prior to the first dose of study treatment or has not recovered from prior surgery.
4. Has traditional Chinese medicine or Chinese patent medicine preparation with anti-cancer indication within 2 weeks prior to the first dose of study treatment.
5. Requiring corticosteroids (Prednisone >10 mg/day or equivalent analogue) or other immunosuppressive agents within 2 weeks prior to the first dose of study treatment. 6. Patients without active autoimmune disease using inhaled prednisone >10 mg/day will not be excluded from the study.

7. Has a history of organ transplantation or required long-term treatment with corticosteroids.

8. Hypothyroidism, hypoadrenalism or hypopituitarism that can be controlled only with hormone replacement therapy, type I diabetes, psoriasis or leucoderma not requiring systematic treatment.

9. Not recovered from the toxicity of prior anti-cancer therapy, i.e., not recovered to baseline, Grade 0-1 (NCI-CTCAE 5.0, except alopecia) or per inclusion/exclusion criteria in protocol. Under rational expectation, irreversible toxicities (e.g., hearing loss) which will not be worsened by study treatments may be enrolled in the study.

10. Has an additional malignancy that has progressed or required treatment within 5 years prior to randomization (basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ such as breast cancer, prostate cancer are acceptable if they have undergone potentially curative therapy；Remarks: Localized low-risk prostate cancer [ patietns with stage ≤ T2a, Gleason score ≤ 6 and PSA < 10ng/mL at the time of diagnosis (as measured) can be included in this study if the subject has received radical therapy and has no evidence for biochemical recurrence(PROSTATE specific antigen,PSA)].

11. Has a history of active central nervous system (CNS) metastasis or CNS metastasis had been confirmed by radiological examination (MRI or CT) at baseline within 30 days prior to the first dose of study drug. Subjects may participate who had been stable at least for 3 months after prior surgery or RT for brain or meningeal metastasis and discontinued systemic treatment with corticosteroids (Prednisone >10 mg/day or equivalent analogue) for at least 4weeks. Subjects may participate in the study if their CNS metastases are adequately treated to meet the requirements specified in the inclusion criteria, and their neurological symptoms recover to grade 0-1 (CTCAE 5.0) for at least 2 weeks prior to inclusion (except for residual signs or symptoms associated with CNS treatment).

12. Poorly controlled hypertension (systolic blood pressure ≥ 150mmHg and/or diastolic blood pressure ≥ 90mmHg).

13. Presence of the following cardiovascular events within 6 months prior to randomization: Myocardial infarction Unstable angina pectoris Cardiac angioplasty or stent Coronary/peripheral artery bypass graft Grade III or IV congestive heart failure per New York Heart Association Cerebrovascular accident or transient ischemic attack QT interval (QTc) ≥ 480 msec corrected with heart rate (Bazett's formula); 14. Has active hemorrhage or history of other significant hemorrhage episodes within 30 days prior to randomization.

15. Has deep vein thrombosis or pulmonary embolism within 6 months prior to randomization.

16. Has arterial thrombosis within 12 months prior to randomization. 17. Has clinically significant gastrointestinal (GI) abnormalities including: Malabsorption, total gastrectomy or any other condition that might affect the absorption of orally taken medication.

Active ulcer under treatment in the past 6 months; Active GI bleeding (e.g., hematemesis, hematochezia or melena) in the past 3 months, and without evidence of resolution documented by endoscopy or colonoscopy.

Intraluminal metastatic lesion with suspected hemorrhage, inflammatory bowel disease, ulcerative colitis, GI perforation, or other GI conditions associated with increased risk of perforation.

18. Has a history of or current (non-infective) pneumonia/ interstitial lung disease that required steroids.

19. Has an active infection requiring systemic therapy. Has a known history of Human Immunodeficiency Virus (HIV) infection (HIV antibody positive), HBV or HCV infection (Patients with positive HBsAg or negative HBsAg, but positive HBcAb will be enrolled in the study when HBV DNA was tested in central laboratory and lower than ULN. Patients with a history of HCV infection may participate in the study if the result of HCV RNA test was negative during screening period).

20. Has received a live virus vaccine within 30 days prior to randomization, including (but not limited to) mumps, rubella, measles, varicella/ herpes zoster (chicken pox), yellow fever, rabies, Bacille Calmette-Guérin (BCG) and typhoid vaccine. Inactivated virus vaccines are allowed.

21. Has a history of hypersensitivity reaction, including (but not limited to) antibodies and TKIs.

22. Known history of psychiatric disorders or drug abuse. 23. Has evidence of inadequate wound healing. 24. Has current use (within 7 days of randomization) or anticipated need for treatment drugs what are known strong CYP3A4/5 inhibitor and CYP3A4/5 inducer (including, but not limited to, carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin and St. John's wort) or the drugs that are known with proarrhythmic potential (including, but not limited to, terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol and benazapril, etc.).

25. Has a history or current evidence on any condition, therapy or laboratory abnormality that might confound the results of the study, interfere with subject's participation for the full duration of the study, or is not in the best interest of subject to participate, in the opinion of investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
ORR assessed by investigators per RECIST 1.1 | Up to approximately 2 years
  The treatment effect of with ICI plus axitinib will be assessed using RECIST 1.1 to determine tumor response.

SECONDARY OUTCOMES:
PFS assessed by investigators per RECIST 1.1 | Up to approximately 2 years
  The treatment effect of with ICI plus axitinib will be assessed using RECIST 1.1 to determine tumor response.

CONTACTS AND LOCATIONS:
Overall Officials: Xinan Sheng, MD., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (2):
- China (2):
  - Department of Genitourinary Oncology, Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No